CLINICAL TRIAL: NCT01852045
Title: BOTOX® in the Treatment of Urinary Incontinence Due to Neurogenic Detrusor Overactivity in Patients 5 to 17 Years of Age
Brief Title: Study of OnabotulinumtoxinA (BOTOX®) for Urinary Incontinence Due to Neurogenic Detrusor Overactivity in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-120; 2012-004877-26 (EudraCT Number)
Record Dates: First submitted 2013-05-09; First posted 2013-05-13 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OnabotulinumtoxinA 50 U (Experimental): OnabotulinumtoxinA (botulinum toxin Type A) 50 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1. Participants were eligible for retreatment in study 191622-121 (NCT01852058) if qualified.
  Interventions: Biological: OnabotulinumtoxinA
- OnabotulinumtoxinA 100 U (Experimental): OnabotulinumtoxinA (botulinum toxin Type A) 100 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1. Participants were eligible for retreatment in study 191622-121 if qualified.
  Interventions: Biological: OnabotulinumtoxinA
- OnabotulinumtoxinA 200 U (Experimental): OnabotulinumtoxinA (botulinum toxin Type A) 200 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1. Participants were eligible for retreatment in study 191622-121 if qualified.
  Interventions: Biological: OnabotulinumtoxinA

INTERVENTIONS:
Biological: OnabotulinumtoxinA — OnabotulinumtoxinA injected into the detrusor wall on Day 1.
  Other Names: BOTOX®; botulinum toxin Type A

SUMMARY:
This study will evaluate the 3 doses of onabotulinumtoxinA (botulinum toxin Type A) for the treatment of urinary incontinence due to neurogenic detrusor overactivity in pediatric participants between the ages of 5 to 17 years to determine if 1 or more doses were safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence due to neurogenic detrusor overactivity
* Regularly using clean intermittent catheterization to empty the bladder

Exclusion Criteria:

* Surgery of the spinal cord within 6 months
* Diagnosis of cerebral palsy
* Current or planned use of a baclofen pump
* Current or planned use of an electrostimulation/neuromodulation device for urinary incontinence
* Use of an indwelling catheter for urinary incontinence instead of using clean intermittent catheterization to empty the bladder
* Previous or current use of botulinum toxin therapy of any serotype for any urological condition, or treatment with botulinum toxin of any serotype within 3 months for any other condition or use
* Myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Furmanov, Study Director — Allergan
Locations (31):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - William Beaumont Hospital Research Institute, Royal Oak, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Pediatric Urology Associates, PC, Tarrytown, New York
  - McKay Urology Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oklahoma Childrens Hospital, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - UZ Antwerpen, Antwerp
  - UZ Gent , Urology, Ghent
  - UZ Leuven, Leuven
- Canada (2):
  - McMaster University Medical Centre, Hamilton, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
- France (4):
  - Hopital Pellegrin - Enfants, Bordeaux
  - CHU de Limoges - Hopital Mere et l'Enfant, Limoges
  - Hopital Trousseau, Paris
  - Necker Enfants Malades Hospital, Paris
- Italy (2):
  - Seconda Università di Napoli, Caserta
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
- Poland (3):
  - Copernicus Podmiot Leczniczy Sp. z o. o., Kliniczny Oddzial Chirurgii i Urologii Dzieci i Mlodziezy GUMed, Gdansk
  - Specjalistyczny Gabinet Lekarski, Poznan
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw
- Ankara University Medical Faculty Cebeci Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 114 patients were enrolled and randomized into the study; 113 received study treatment.
Groups:
- OnabotulinumtoxinA 100 U: OnabotulinumtoxinA 100 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1. Participants were eligible for retreatment in study 191622-121 if qualified.
- OnabotulinumtoxinA 200 U: OnabotulinumtoxinA 200 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1. Participants were eligible for retreatment in study 191622-121 if qualified.
Period: Overall Study
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Started | 39 | 45 | 30
mITT Population | 38 | 45 | 30
Safety Population | 38 | 45 | 30
Completed | 33 | 41 | 26
Not Completed | 6 | 4 | 4
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Other Miscellaneous Reasons | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U | Total
Number analyzed (Participants) | 39 | 45 | 30 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (3.45) | 10.8 (3.26) | 11.9 (3.13) | 11.3 (3.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 15 | 49
  Male | 20 | 30 | 15 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 34 | 22 | 85
  Black or African American | 6 | 3 | 2 | 11
  Asian | 1 | 2 | 1 | 4
  Hispanic | 1 | 3 | 3 | 7
  Other | 2 | 3 | 2 | 7
Daily Daytime Average Frequency of Urinary Incontinence Episodes [Mean (Full Range); unit: urinary incontinence episodes per day] — Urinary incontinence was defined as involuntary loss of urine as recorded by the participant in a bladder diary during the 2 consecutive days (normalized to a 12-hour daytime period) prior to the study visit. Daytime was defined as the time between waking up to start the day and first morning catheterization and going to bed to sleep for the night. The number of incontinence episodes were averaged daily during this period. Population: Modified Intent-to-Treat (mITT) population included participants who received study drug on Day 1, analyzed on as-randomized basis, except those who received less than their randomized dose due to weight and dose limit of 6 U/kg, allocated to nearest dose group based on dose received.
  urinary incontinence episodes per day
    number analyzed (Participants) | 38 | 45 | 30 | 113
    (all) | 2.81 [0.8 to 6.7] | 2.99 [1.3 to 6.1] | 3.68 [0.5 to 29.5] | 3.16 [0.5 to 29.5]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Average Frequency of Daytime Urinary Incontinence Episodes
Description: Urinary incontinence was defined as involuntary loss of urine as recorded by the participant in a bladder diary during the 2 consecutive days (normalized to a 12-hour daytime period) prior to the study visit. Daytime was defined as the time between waking up to start the day and first morning catheterization and going to bed to sleep for the night. The number of incontinence episodes were averaged daily during this period. A negative change from Baseline indicates improvement. Least squares estimates were based on an Analysis of Covariance (ANCOVA) model.
Time Frame: Baseline (Day -28 to Day -1) to 2 consecutive days prior to Week 6
Population: mITT population included participants who received study drug on Day 1, analyzed on as-randomized basis, except those who received less than their randomized dose due to weight and dose limit of 6 U/kg, allocated to nearest dose group based on dose received. Missing data are imputed up to Week 6 using Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: urinary incontinence episodes per day
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 38 | 45 | 30
urinary incontinence episodes per day | -1.30 (0.205) | -1.30 (0.189) | -1.34 (0.245)
Statistical Analysis 1: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 100 U; Test type: Superiority; p = 0.9949, ANCOVA; Least Squares Mean Difference = 0.00, 95% CI 2-sided [-0.549 to 0.545], Standard Error of Mean 0.276 — Least squares estimates and contrast t-test were based on ANCOVA model with baseline value as covariate and treatment group, age, baseline daytime urinary incontinence episodes, anticholinergic therapy at baseline as factors
Statistical Analysis 2: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 200 U; Test type: Superiority; p = 0.9123, ANCOVA; Least Squares Mean Difference = -0.04, 95% CI 2-sided [-0.673 to 0.602], Standard Error of Mean 0.321 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is defined as any new adverse event or worsening of an existing condition after initiation of treatment.
Time Frame: First study treatment to 12 weeks after last treatment (Up to 48 weeks after first study injection)
Population: Safety population included participants who underwent treatment procedure and received study drug on randomization/Day 1, except those who received less dose due to 6 U/kg weight cap, were allocated to nearest dose group based on the actual dose received.
Measure: Count of Participants; unit: Participants
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 38 | 45 | 30
Participants | 27 | 33 | 23

3. Secondary Outcome: Change From Baseline in Average Urine Volume at First Morning Catheterization
Description: The change in urine volume at first morning catherization was recorded by the participant in a bladder diary in the 2 consecutive days during the week prior to the study visit. A positive change from Baseline indicates improvement. Least squares estimates were based on an ANCOVA model.
Time Frame: Baseline (Day -28 to Day -1) to 2 consecutive days prior to Week 6
Population: mITT population included participants who received study drug on Day 1, analyzed on as-randomized basis, except those who received less than their randomized dose due to weight and dose limit of 6 U/kg, allocated to nearest dose group based on dose received. Number analyzed is number of participants with non-missing values at the specified Visit.
Measure: Least Squares Mean (Standard Error); unit: milliliters (mL)
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 36 | 43 | 27
milliliters (mL) | 21.93 (14.676) | 34.90 (13.580) | 87.49 (17.808)
Statistical Analysis 1: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 100 U; Test type: Superiority; p = 0.5117, ANCOVA; Least Squares Mean Difference = 12.97, 95% CI 2-sided [-26.120 to 52.064], Standard Error of Mean 19.694 — Least squares estimates and contrast t-test are based on ANCOVA model with baseline value as covariate and treatment group, age, baseline daytime urinary incontinence episodes, anticholinergic therapy at baseline as factors
Statistical Analysis 2: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 200 U; Test type: Superiority; p = 0.0055, ANCOVA; Least Squares Mean Difference = 65.57, 95% CI 2-sided [19.711 to 111.421], Standard Error of Mean 23.101 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Percentage of Participants With Night Time Urinary Incontinence
Description: Urinary incontinence was defined as involuntary loss of urine and the presence or absence of night time urinary incontinence was recorded by the participant in a bladder diary in the 2 consecutive days (normalized to a 12-hour daytime period) during the week prior to the study visit. Night time was defined as the time between going to bed to sleep for the night and waking up to start the day. The percentage of participants with night time urinary incontinence is presented in categories (0, 1, 2 nights).
Time Frame: Baseline (Day -28 to Day -1), Week 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 38 | 45 | 28
percentage of participants
  Baseline (BL): 0 nights of incontinence | 0.0 | 13.3 | 3.6
  BL: 1 night of incontinence | 13.2 | 2.2 | 14.3
  BL: 2 nights of incontinence | 86.8 | 84.4 | 82.1
  Week 6: 0 nights of incontinence: number analyzed (Participants) | 36 | 43 | 28
  Week 6: 0 nights of incontinence | 30.6 | 32.6 | 28.6
  Week 6: 1 night of incontinence: number analyzed (Participants) | 36 | 43 | 28
  Week 6: 1 night of incontinence | 16.7 | 16.3 | 28.6
  Week 6: 2 nights of incontinence: number analyzed (Participants) | 36 | 43 | 28
  Week 6: 2 nights of incontinence | 52.8 | 51.2 | 42.9

5. Secondary Outcome: Change From Baseline in Maximum Cystometric Capacity (MCC)
Description: The MCC was defined by urodynamics, as the volume infused before the participant felt they could no longer delay micturition (has a strong desire to void), had a leakage, or 500 mL was instilled. A positive change from Baseline indicates improvement (increase) in the maximum volume of urine the bladder holds. Least squares estimates were based on an ANCOVA model.
Time Frame: Baseline (Day -28 to Day -1) to Week 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 34 | 38 | 28
mL | 62.06 (14.339) | 48.57 (13.549) | 63.55 (17.363)
Statistical Analysis 1: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 100 U; Test type: Superiority; p = 0.4948, ANCOVA; Least Squares Mean Difference = -13.49, 95% CI 2-sided [-52.605 to 25.626], Standard Error of Mean 19.673 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 200 U; Test type: Superiority; p = 0.9471, ANCOVA; Least Squares Mean Difference = 1.49, 95% CI 2-sided [-43.012 to 45.991], Standard Error of Mean 22.382 — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Percentage of Participants With Involuntary Detrusor Contractions (IDC)
Description: Urodynamic tests were performed by site personnel qualified for performing pressure/flow cystometry. The results were verified by an independent central reviewer. Cystometry was used to measures the presence of involuntary detrusor contractions upon filling. A reduction in IDCs from Baseline to Week 6 indicates improvement.
Time Frame: Baseline (Day -28 to -1) and Week 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 38 | 45 | 30
percentage of participants
  Baseline: number analyzed (Participants) | 36 | 42 | 27
  Baseline | 94.4 [81.34 to 99.32] | 88.1 [74.37 to 96.02] | 92.6 [75.71 to 99.09]
  Week 6: number analyzed (Participants) | 34 | 38 | 28
  Week 6 | 61.8 [43.56 to 77.83] | 44.7 [28.62 to 61.70] | 46.4 [27.51 to 66.13]
Statistical Analysis 1: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 100 U; Week 6; Test type: Superiority; p = 0.2027, Cochran-Mantel-Haenszel — P-values for pairwise comparisons are obtained from 2-sided CMH test, stratified by age (<12 years or >=12 years), baseline daytime urinary incontinence episodes (<=6 or >6) and anticholinergic therapy (yes/no); Relative Risk = 0.7, 95% CI 2-sided [0.45 to 1.14]
Statistical Analysis 2: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 200 U; Week 6; Test type: Superiority; p = 0.1564, Cochran-Mantel-Haenszel — P-values for pairwise comparisons are obtained from a 2-sided CMH test, stratified by age (< 12 years or >= 12 years), baseline daytime urinary incontinence episodes (<= 6 or > 6) and anticholinergic therapy (yes/no); Relative Risk = 0.8, 95% CI 2-sided [0.40 to 1.21]

7. Secondary Outcome: Change From Baseline in Maximum Detrusor Pressure During the First IDC (PdetMax1stIDC) in Participants With IDC
Description: Urodynamic tests were performed by site personnel qualified for performing pressure/flow cystometry. The results were verified by an independent central reviewer. Cystometry was used to measures the pressure inside of the bladder to see how well the bladder was working. A negative change from Baseline indicates improvement. Least squares estimates were based on an ANCOVA model.
Time Frame: Baseline (Day-28 to Day-1) to Week 6
Population: mITT population included participants who received study drug on Day 1, analyzed on as-randomized basis, except those who received less than their randomized dose due to weight and dose limit of 6 U/kg, allocated to nearest dose group based on dose received. Only participants who experienced an IDC are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: centimeters of water (cm H2O)
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 21 | 17 | 12
centimeters of water (cm H2O) | -7.64 (5.301) | -12.13 (5.573) | -5.46 (8.267)
Statistical Analysis 1: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 100 U; Test type: Superiority; p = 0.5524, ANCOVA; Least Squares Mean Difference = -4.49, 95% CI 2-sided [-19.648 to 10.669], Standard Error of Mean 7.488 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 200 U; Test type: Superiority; p = 0.8313, ANCOVA; Least Squares Mean Difference = 2.18, 95% CI 2-sided [-18.427 to 22.795], Standard Error of Mean 10.181 — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Change From Baseline in Maximum Detrusor Pressure (PdetMax) During the Storage Phase
Description: as for outcome 7
Time Frame: Baseline (Day 1) to Week 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: cm H2O
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 34 | 38 | 28
cm H2O | -12.88 (3.793) | -20.09 (3.632) | -27.31 (4.557)
Statistical Analysis 1: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 100 U; Test type: Superiority; p = 0.1737, ANCOVA; Least Squares Mean Difference = -7.21, 95% CI 2-sided [-17.653 to 3.238], Standard Error of Mean 5.253 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: OnabotulinumtoxinA 50 U vs OnabotulinumtoxinA 200 U; Test type: Superiority; p = 0.0157, ANCOVA; Least Squares Mean Difference = -14.43, 95% CI 2-sided [-26.061 to -2.793], Standard Error of Mean 5.850 — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Change From Baseline in Detrusor Leak Point Pressure (DLPP) During the Storage Phase
Description: DLPP was defined as the lowest detrusor pressure at which urine leakage occurs in the absence of either a detrusor contraction or increased intra-abdominal pressure. Urodynamic tests were performed by site personnel qualified for performing pressure/flow cystometry. The results were verified by an independent central reviewer. Cystometry was used to measures the pressure inside of the bladder to see how well the bladder was working. A negative change from Baseline indicates improvement. Least squares estimates are based on an ANCOVA model.
Time Frame: Baseline (Day -28 to -1) to Week 6
Population: mITT population included participants who received study drug on Day 1, analyzed on as-randomized basis, except those who received less than their randomized dose due to weight and dose limit of 6 U/kg, allocated to nearest dose group based on dose received. Only participants who experienced a leak during urodynamics are included in the analysis.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 2 | 1 | 1
cm H2O | 9.50 (2.121) | -39.00 (0.000) | 12.00 (0.000)

10. Secondary Outcome: Time to Participant Request for Retreatment
Description: Time from treatment on Day 1 to request for retreatment was estimated. For those participants who did not request retreatment, their data was censored using the date of their last study visit.
Time Frame: 48 weeks
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 27 | 35 | 23
weeks | 30.6 [23.10 to 39.10] | 24.1 [18.10 to 27.60] | 29.6 [16.30 to 37.30]

11. Secondary Outcome: Time to Participant Qualification for Retreatment
Description: In order to qualify for retreatment, the criteria listed below must be fulfilled at the qualification for retreatment visit: Participant/parent/caregiver requests retreatment, participant has a total of at least 2 daytime urinary incontinence episodes over the 2-day bladder diary collection period, at least 12 weeks has elapsed since treatment 1 and participant has not experienced a serious treatment-related adverse event at any time.
Time Frame: 48 weeks
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 27 | 35 | 23
weeks | 35.0 [23.10 to 39.10] | 25.0 [20.00 to 32.10] | 29.6 [16.30 to 38.00]

ADVERSE EVENTS:
Time Frame: First study treatment to 12 weeks after last treatment (Up to 48 weeks after first study injection)
Description: Safety population included participants who underwent treatment procedure and received study drug on randomization/Day 1, except those who received less dose due to 6 U/kg weight cap, were allocated to nearest dose group based on the actual dose received.
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/45 | 0/30
Serious Adverse Events (participants affected / at risk) | 4/38 | 3/45 | 2/30
Other Adverse Events (participants affected / at risk) | 27/38 | 33/45 | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA 50 U (N=38) | OnabotulinumtoxinA 100 U (N=45) | OnabotulinumtoxinA 200 U (N=30)
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Encephalitis viral (Infections and infestations) | 0 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA 50 U (N=38) | OnabotulinumtoxinA 100 U (N=45) | OnabotulinumtoxinA 200 U (N=30)
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Pyrexia (General disorders) | 2 | 4 | 0
Suprapubic pain (General disorders) | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 9 | 13 | 7
Bacteriuria (Infections and infestations) | 6 | 7 | 6
Pharyngitis (Infections and infestations) | 3 | 3 | 0
Gastroenteritis (Infections and infestations) | 2 | 3 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 2
Headache (Nervous system disorders) | 1 | 7 | 2
Leukocyturia (Renal and urinary disorders) | 1 | 3 | 4
Hydronephrosis (Renal and urinary disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT01852045/SAP_000.pdf
  • Study Protocol (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT01852045/Prot_001.pdf